CLINICAL TRIAL: NCT02088502
Title: Comparative Evaluation of the Effect of Theophylline Plus N-acetylcysteine, Theophylline Alone, and N-acetylcysteine Alone in Preventing Contrast-induced Nephropathy in Patients With Moderate to High Risk Undergoing Coronary Angiographic Procedures
Brief Title: Theophylline, N-acetylcysteine, and Theophylline Plus N-acetylcysteine in Preventing Contrast-induced Nephropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mortaza Arabmomeni, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 392300
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Contrast-Induced Nephropathy
Keywords: Coronary Angiography; Side Effects; Contrast-Induced Nephropathy; Prevention
MeSH Terms: interventions — Acetylcysteine; Theophylline; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- N-acetylcysteine (Active Comparator): Patients in the N-acetylcysteine group receive 600 mg non-effervescent N-acetylcysteine tablet plus placebo twice daily from 24 hours before to 48 hours after administration of contrast material.
  Interventions: Drug: N-acetylcysteine; Drug: 0.9% sodium chloride
- Theophylline (Active Comparator): Patients in the Theophylline group receive 200 mg Theophylline slow-release tablet plus placebo twice daily from 24 hours before to 48 hours after administration of contrast material.
  Interventions: Drug: Theophylline; Drug: 0.9% sodium chloride
- Theophylline plus N-acetylcysteine (Active Comparator): Patients in the Theophylline plus N-acetylcysteine group receive Theophylline slow-release 200 mg tablet plus non-effervescent N-acetylcysteine 600 mg tablet twice daily from 24 hours before to 48 hours after administration of contrast material.
  Interventions: Drug: N-acetylcysteine; Drug: Theophylline; Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: N-acetylcysteine
  Arms: N-acetylcysteine; Theophylline plus N-acetylcysteine
Drug: Theophylline
  Arms: Theophylline; Theophylline plus N-acetylcysteine
Drug: 0.9% sodium chloride — All patients are hydrated with 0.9% sodium chloride (1 mL/kg/hour) for 24 hours, 12 hours before operation. Patients with left ventricular ejection fraction less than 40% or New York Heart Association functional class III-IV, are hydrated with 0.5 mL/kg per hour.

SUMMARY:
The aim of this study is to determine the efficacy of Theophylline, N-Acetylcysteine and, and Theophylline plus N-acetylcysteine in the prevention of contrast-induced nephropathy. Investigators assume that Theophylline plus N-acetylcysteine is more effective than Theophylline alone and N-acetylcysteine alone. Investigators include patients referring for elective coronary angiography or angioplasty and allocate them to each of the mentioned treatments from 24 hours before to 48 hours after administration of contrast material. Investigators then measure serum creatinine and see if it is raised by ≥ 0.5 mg/dL or ≥ 25% of the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* candidate of elective coronary angiography or angioplasty
* at least moderate risk for contrast induced nephropathy

Exclusion Criteria:

* unstable angina or myocardial infarction, cardiac arrhythmia, seizures, acute renal failure, end-stage renal disease
* unstable serum creatinine
* unstable hemodynamic
* intravascular administration of contrast material in the past month
* using theophylline or N-acetylcysteine in the past month,
* known hypersensitivity to theophylline or N-acetylcysteine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Plasma creatinine level | up to 48h after contrast injection
  Plasma creatinine level is measured at baseline and after 48 hours of contrast injection. Increase in plasma creatinine level ≥ 0.5 mg/dL or ≥ 25% of the baseline creatinine after 48 hours of contrast injection will be considered contrast induced nephropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Mortaza Arabmomeni, M.D., Study Director — Isfahan University of Medical Sciences
Locations (1):
- Chamran Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Albabtain MA, Almasood A, Alshurafah H, Alamri H, Tamim H. Efficacy of ascorbic acid, N-acetylcysteine, or combination of both on top of saline hydration versus saline hydration alone on prevention of contrast-Induced nephropathy: a prospective randomized study. J Interv Cardiol. 2013 Feb;26(1):90-6. doi: 10.1111/j.1540-8183.2012.00767.x. Epub 2012 Sep 20. PMID 22994682